CLINICAL TRIAL: NCT06983353
Title: Evaluation of Transphyseal Screw Guided Growth Technique for Correction of Coxa Valga in Cerebral Palsy Children With Hip Sublaxation A Pilot Study
Brief Title: Guided Growth Technique Use In Treatment Of Hip Sublaxation In CP Childern
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Adel Fathy Abdel aleem (Other)
Responsible Party: Sponsor-Investigator, Mohamed Adel Fathy Abdel aleem, doctor, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: guided growth in cp childern
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy (CP); Guided Growth
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: transphyseal screw — transphyseal screw in proximal femoral physis

SUMMARY:
To evaluate the change in femoral neck-shaft angle (coxa valga) following transphyseal screw insertion in children with CP.

DETAILED DESCRIPTION:
The hip is one of the most common involved joint in cerebral palsy. Hip displacement occurs in more than 33% of children with cerebral palsy, with a higher prevalence in nonambulatory children. Hip displacement in this population is typically progressive. Hip dislocation can result in pain and difficulty with sitting and perineal care. Hip Surveillance in Children with Cerebral Palsy.

Traditional surgical management, typically reserved for hips with a migration percentage of 40% or more, includes hip reconstruction involving soft tissue releases, femoral and pelvic osteotomies. These procedures are associated with significant perioperative morbidity, including pain; increased blood loss; and lengthy anesthetic and inpatient recovery times, often complicated with peri-operative infections. With improved surgical techniques, orthopedic implants and enhanced postoperative pathways, weightbearing can be resumed shortly after surgery; however, traditional treatment commonly included a period of non-weight-bearing, with some surgeons preferring to augment their reconstruction with a hip spica or abduction brace .

Guided growth procedures are well established in the treatment for the gradual correction of angular and rotational limb deformities in children. Anterior hemiepiphysiodesis of the distal femur has been shown to be effective in the treatment of fixed flexion deformity of the knee when compared to traditional osteotomies. shows intra-operative radiographs of this minimally invasive technique, which has been recently applied to the proximal femoral physis for various conditions. By placing a screw over the physis on the medial side, the tethering that occurs on the medial side will result in progressive varus of the proximal femur. It is understood that this manipulation of the proximal femoral anatomy can alter the course of secondary acetabular dysplasia .Furthermore, it is recognized that guided growth procedures of the proximal femoral physis can be carried out as day case procedures, require a shorter operating time and allow for immediate weight bearing/standing when performed in non-ambulatory patients.

Type of the study: Prospective cohort study Study Setting: Assiut University Hospitals, Department of Orthopaedics and Traumatology

Preoperative assessment :

A-Clinical for GMFCS B- Radiological AP and Lateral pelvis for the migration percentage (MP), head/neck-shaft angle (HSA/NSA) and acetabular index (AI) Procedure: Insertion of a transphyseal fully threaded cannulated screw at proper size across the infromedial proximal femoral physis under fluoroscopic guidance +/- soft tissue release , Abductor brace , hip spicca , and ankle foot orthosis .

* Postoperative Care:
* Weight-bearing as tolerated.
* Physical therapy to improve hip abductor strength and range of motion.
* Regular follow-up at 1.5, 3, 6, 12, and 24 months and uptill .

ELIGIBILITY:
Inclusion Criteria:

* children aged 3-12 yrs diagnosed with CP ( GMFCS level l_lV )
* Neck-Shaft angle >150
* early hip sub laxation ( migration percentage < 50% )

Exclusion Criteria:

* Sever hip sub laxation ( migration percentage> 50 % )
* Children below 3 yrs and above 12
* Pathological bone
* medical contraindications to surgery

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in femoral neck-shaft angle (measured on anteroposterior pelvic radiographs). | - Regular follow-up at 1.5, 3, 6, 12, and 24 months .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Background] Hsieh HC, Wang TM, Kuo KN, Huang SC, Wu KW. Guided Growth Improves Coxa Valga and Hip Subluxation in Children with Cerebral Palsy. Clin Orthop Relat Res. 2019 Nov;477(11):2568-2576. doi: 10.1097/CORR.0000000000000903. PMID 31425278
- [Background] Lebe M, van Stralen RA, Buddhdev P. Guided Growth of the Proximal Femur for the Management of the 'Hip at Risk' in Children with Cerebral Palsy-A Systematic Review. Children (Basel). 2022 Apr 25;9(5):609. doi: 10.3390/children9050609. PMID 35626786